CLINICAL TRIAL: NCT03217201
Title: Systematic Light Exposure to Treat Cancer-Related Fatigue in Breast Cancer Patients
Brief Title: Systematic Light Exposure for Fatigue in Breast Cancer Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Icahn School of Medicine at Mount Sinai (Other)
Collaborators: Memorial Sloan Kettering Cancer Center (Other); National Cancer Institute (NCI) (NIH); City of Hope Medical Center (Other)
Responsible Party: Principal Investigator, William H. Redd, Professor, Icahn School of Medicine at Mount Sinai
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: GCO 15-1783; 1R01CA207446-01A1 (NIH)
Record Dates: First submitted 2017-07-11; First posted 2017-07-14 (Actual); Last update posted 2023-08-23 (Actual); Status verified 2023-08

CONDITIONS: Cancer-related Problem/Condition; Fatigue; Circadian Rhythm Disorders
Keywords: Breast Cancer; Oncology; Circadian Rhythm; Light Therapy; Chemotherapy side effects
MeSH Terms: conditions — Fatigue; Chronobiology Disorders; Breast Neoplasms; Neoplasms

STUDY DESIGN:
Intervention Model Description: Stratified by adjuvant and neoadjuvant chemotherapy treatments, then randomly assigned to one of two light treatment conditions.
Who Masked: Participant
Masking Description: The participant does not know his or her study condition.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Adjuvant, Experimental Light (Experimental): 30 minutes of experimental systematic light exposure daily for duration of chemotherapy treatment.
  Interventions: Device: Light Glasses (Experimental)
- Adjuvant, Comparison Light (Active Comparator): 30 minutes of comparison systematic light exposure daily for duration of chemotherapy treatment.
  Interventions: Device: Light Glasses (Comparison)
- Neo-Adjuvant, Experimental Light (Experimental): 30 minutes of experimental systematic light exposure daily for duration of chemotherapy treatment.
  Interventions: Device: Light Glasses (Experimental)
- Neo-Adjuvant, Comparison Light (Active Comparator): 30 minutes of comparison systematic light exposure daily for duration of chemotherapy treatment.
  Interventions: Device: Light Glasses (Comparison)

INTERVENTIONS:
Device: Light Glasses (Experimental) — The light glasses emit light from LEDs at a distance of 15 millimeters (15mm, 0.015.) from the eye. The device Is classified as safe for the eyes in accordance with the international standard IEC 62471 and complies with the United States of America's FCC marking, and is designed to be worn on the participant's head, similarly to a pair of glasses. For safety purposes, the light glasses do not contain UV or infra-red light.
  Arms: Adjuvant, Experimental Light; Neo-Adjuvant, Experimental Light
Device: Light Glasses (Comparison) — The light glasses emit light from LEDs at a distance of 15 millimeters (15mm, 0.015.) from the eye. The device Is classified as safe for the eyes in accordance with the international standard IEC 62471 and complies with the United States of America's FCC marking, and is designed to be worn on the participant's head, similarly to a pair of glasses. For safety purposes, the light glasses do not contain UV or infra-red light.
  Arms: Adjuvant, Comparison Light; Neo-Adjuvant, Comparison Light

SUMMARY:
Cancer related fatigue (CRF) is a stressful and constant tiredness related to cancer and/or its treatment. CRF is the most intense during treatment and can severely interfere with activities of daily living, such as tasks that require physical strength or thinking clearly. Prevalence of CRF has been reported to be as high as 94% during chemotherapy and as high as 34% five years after completion of treatment (Rotonda et al. 2013; Minton & Stone 2008). There is currently no generally-accepted treatment for CRF. However, there is evidence to suggest that light therapy can help with CRF. Non-pharmacological interventions for CRF have also been studied but are costly to implement and involve significant patient burden, particularly among those in active treatment. Given the clinical impact of CRF, the goal of this project is to investigate a novel, low-cost and low-burden intervention for Breast Cancer patients using a particular kind of light treatment called systematic light exposure (sLE) to treat CRF. Two hundred forty-eight breast cancer (BC) patients undergoing adjuvant or neoadjuvant chemotherapy will be recruited from Memorial Sloan Kettering Cancer Center, and City of Hope. The light will be administered by light glasses daily throughout entire duration of chemotherapy. Outcomes will be assessed at eight timepoints during chemo, and a series of follow up assessments at 1 week, 1-month, 3-months and 6-months post-chemotherapy. This study will have major public health relevance as it will determine if an easy-to-deliver, inexpensive, and low patient burden intervention effectively reduces CRF or prevents it from worsening during chemotherapy. Specific Aims: Aim 1: Determine if sLE prevents CRF from worsening in BC patients undergoing chemotherapy Aim 2: Determine whether sLE affects sleep, depression and circadian activity rhythms. Exploratory Aim 3: Investigate sLE normalizes circadian cortisol rhythms. Exploratory Aim 4: Examine whether the effects of sLE on fatigue are moderated/mediated by sleep quality, depression, and/or circadian rhythms.

ELIGIBILITY:
Inclusion Criteria:

* Newly diagnosed patients with stage 1 through 3a Breast Cancer scheduled to receive a 12-week, 16-week, 18-week, 20-week, or 24-week chemotherapy regimen, adjuvant, neoadjuvant, or already receiving chemotherapy.
* MSH, COH and MSK can recruit participants schedule to go on aromatase inhibitors after treatment.
* Currently over the age of 18.
* English language proficient.
* Able to provide informed consent.

Exclusion Criteria:

* Under age 18
* Breast cancer patients scheduled to undergo chemo regimen other than the 12-week, 18-week, 20-week, or 24-week regimen
* Stage 3B breast cancer inflammatory or Stage 4 breast cancer
* Pregnancy
* Currently employed in night shift work
* Confounding underlying medical illnesses which may cause fatigue (e.g., severe Anemia not controlled by medication, per self-report corroborated by medical chart review (e.g., Hb<10gm/dl))
* Eye Diseases which limit the ability of light to be processed (e.g., untreated cataracts, severe glaucoma, macular degeneration, blindness, pupil dilation problems or retina damage)
* Secondary cancer diagnosis (prior or current) within the past 5 years
* Severe sleep disorders (e.g., Narcolepsy)
* Self- reported history of bipolar disorder or manic episodes (which is a contra-indication for light treatment)
* Severe psychological impairment (e.g., hospitalization for depressive episode in the past 12 months
* Previous use of light therapy to alleviate fatigue or depressive symptoms
* Lives outside of the United States throughout the duration of study

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes
Enrollment: 194 (Actual)
Dates: Start 2018-01-25 (Actual); Primary Completion 2022-01-26 (Actual); Study Completion 2022-01-26 (Actual)

PRIMARY OUTCOMES:
FACIT-Fatigue Scale | up to 6 months
  FACIT-Fatigue Scale - The FACIT-Fatigue scale will be used both for selection of patients into the study and as an outcome measure of fatigue. Smith et al. (1999) report that this 13 item scale has excellent test-retest reliability (r = 0.90) and internal consistency reliability (alpha = 0.93-0.95). In addition, criterion related validity studies using objective measures of physical function as the outcome show that patient reported fatigue based on the FACIT- Fatigue can predict these objective measures. This measure is the main tool for measuring fatigue in the Patient-Reported Outcomes Measurement Information System (PROMIS) initiative. Cella (personal communication) has indicated that a FACIT-Fatigue score equal to or less than 33 constitutes clinically significant fatigue.

SECONDARY OUTCOMES:
The Center for Epidemiological Studies Depression Scale (CES-D) | up to 6 months
  The Center for Epidemiological Studies Depression Scale (CES-D) - This 20 item self-report adult instrument is designed to measure common symptoms of depression that have occurred over the past week such as poor appetite, hopelessness, pessimism, and fatigue. Internal consistency using coefficient alpha is estimated to be 0.85 for the general, healthy population, and 0.90 among depressed patient samples.
The Pittsburgh Sleep Quality Index | up to 6 months
  The Pittsburgh Sleep Quality Index consists of 19 self-rated items. Scale reliability is excellent using both an internal consistency criterion (Cronbach's alpha = 0.83) and test-retest reliability (r = 0.85). The validity of the instrument is based on its ability to discriminate patients (those having either sleep problems and/or depressive symptoms) from controls (healthy participants without sleep complaints).
Chronotype (MEQ) | up to 6 months
  The study team will collect data on baseline circadian predispositions using the Morningness-Eveningness Questionnaire, a 19-item self-rated survey designed to measure whether a person's peak alertness is in the morning or the evening. Takes approximately 2 minutes to complete.
Credibility/Expectancy Questionnaire | up to 6 months
  This questionnaire will ask the patient to report whether the patient feels the light box is a useful treatment for CRF. Patient Assessment of Own Functioning Inventory (PAOFI) a 33-item self- report measure of a patient's self-perceptions regarding their functioning in everyday tasks and activities.

CONTACTS AND LOCATIONS:
Overall Officials: William H. Redd, Ph.D., Principal Investigator — Icahn School of Medicine at Mount Sinai
Locations (3):
- United States (3):
  - City of Hope Cancer Center, Duarte, California
  - Icahn School of Medicine at Mount Sinai, New York, New York
  - Memorial Sloan-Kettering Cancer Center, New York, New York

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Rotonda C, Guillemin F, Bonnetain F, Velten M, Conroy T. Factors associated with fatigue after surgery in women with early-stage invasive breast cancer. Oncologist. 2013;18(4):467-75. doi: 10.1634/theoncologist.2012-0300. Epub 2013 Feb 12. PMID 23404818
- [Background] Minton O, Stone P. How common is fatigue in disease-free breast cancer survivors? A systematic review of the literature. Breast Cancer Res Treat. 2008 Nov;112(1):5-13. doi: 10.1007/s10549-007-9831-1. Epub 2007 Dec 7. PMID 18064565
- See also: Breast Cancer — https://www.cancer.org/cancer/breast-cancer.html
- See also: Fatigue — https://medlineplus.gov/fatigue.html
- See also: Cancer-Related Fatigue — https://www.cancer.org/treatment/treatments-and-side-effects/physical-side-effects/fatigue/what-is-cancer-related-fatigue.html